CLINICAL TRIAL: NCT04732897
Title: Impact of a Dynamic Dressing in the Management of Unoperated Hallux Valgus With Theoretical Indication for Surgery: Randomized Open Trial
Brief Title: Impact of a Dynamic Dressing in the Management of Unoperated Hallux Valgus (DYNHALLUX)
Acronym: DYNHALLUX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issue
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-45
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Hallux Abductovalgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Intervention Model Description: Open-label randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): wearing made-to-measure soles with SHORE greater than or equal to 65 (standard of care)
- Interventional arm (Experimental): wearing made-to-measure soles with SHORE greater than or equal to 65 + dynamic dressing of the joint
  Interventions: Procedure: dynamic dressing

INTERVENTIONS:
Procedure: dynamic dressing — Dynamic dressing is made by bandages of the foot with gauze pad, stretchable adhesive tape and elastic compression band
  Arms: Interventional arm

SUMMARY:
Hallux Valgus (HV) is a lateral deviation of the big toe. HV is a deformity of the forefoot centered on the 1st radius (1st metatarsal and big toe). This deformation is characterized by:

* a big toe (hallux) deviated outwards (valgus greater than 12 °)
* a first metatarsal moved medially (varus) (angle M1 / M2> 10 °). We also note the existence of an exostosis formed by the apex of the angle between the 1st metatarsal deviated inwards and the big toe deported outwards. This exostosis corresponds to the head of the 1st metatarsal.

In addition to the pain and the unaesthetic nature induced by this deviation, the modifications of the skeletal axes of the foot cause disorders of its function but also of the joints of the lower limb during standing, walking and running. Axis defects of the lower limbs in varum or valgum also cause deformities in the rearfoot, midfoot and forefoot.

There is no non-surgical curative treatment for this deformity. Different conservative treatment options have been offered for first-line treatment, including different types of physiotherapy, wearing rigid insoles or splints.

Wearing rigid insoles is indicated to "counter" the valgic pressure, thereby reducing pain and high plantar pressure, in patients with HV. Their hardness, expressed in SHORE units, must be greater than 65. By countering the valgic pressure (rearfoot and midfoot), the rigid soles make it possible to contain the development of deformation and stabilize the axis of the first spoke. The speed of hallux deformation is therefore greatly reduced if the soles are worn diligently. But there is little or no impact on the correction of the deformity, but it is stabilized as it is without rapid and major worsening. Indeed, soles with a hardness greater than or equal to 65 SHORE make it possible to avoid the valgum of the hindfoot and midfoot under load and when walking.

Wearing a dynamic splint was studied in a recently published prospective randomized study conducted between 2011 and 2013. This study, concluding that the dynamic splint is not effective in reducing the angle of deformation of the HV, nevertheless shows the reduction in pain during walking and running. The limits of the study lie in the pace of wearing the splint, left to the discretion of patients, during their rest period, and in the duration of the operation, which is not precisely described.

DETAILED DESCRIPTION:
The hypothesis of the study is that a dynamic joint dressing, associated with a rigid orthopedic insole, would make it possible to "reverse" the deformation and re-focus the angles of deformation of the first ray in patients with a HV and already stabilized, i.e. wearer of made-to-measure soles with SHORE greater than or equal to 65 for at least 2 months.

ELIGIBILITY:
Inclusion Criteria:

* hallux valgus on at least one foot theoretically requiring surgical management within 12 months
* reducible hallux valgus
* wearing custom-made orthopedic insoles made by a biomechanical podiatrist - SHORE ≥ 65 - for at least 2 months at the time of inclusion
* beneficiary of a social security scheme
* informed of the study and signed informed consent form

Exclusion Criteria:

* History of hallux valgus correction surgery on the affected foot
* History of traumatic lesion of the M1-P1 metatarsophalangeal joint of the affected foot
* Skin pathology limiting or contraindicating the possibility of dressings according to the judgment of the investigator (eg dyshidrotic eczema, psoriasis or other problematic skin damage located in the foot)
* Acute bursitis
* Clinical and / or radiological stage 1 or more osteoarthritis according to the criteria of Kellgren and Lawrence
* Non-stabilized diabetes and / or diabetes with micro / macrovascular complications
* Patients with neuropathy
* History of gout
* History of rheumatic pathology
* Obliterating arteriopathy of the lower limbs of stage II or more according to the classification of Leriche and Fontaine
* Pregnant woman
* Patients under tutorship or curatorship
* Patients under legal protection
* Patients who do not understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline M1 / P1 angle at day 75 measured by weightbearing foot radiograph | radiograph between day 0 less than 6 months and day 0 and radiograph at day 75
  M1 / P1 angle measured before and after intervention

SECONDARY OUTCOMES:
Variation of the M1 / M2 angle measured by weightbearing foot radiograph | radiograph between day 0 less than 6 months and day 0 and radiograph at day 75
  M1 / M2 angle measured before and after intervention
Variation of the M1 / P1 and M1/M2 angle measured by weightbearing foot radiograph at long time | radiograph at day 75 and at month 6 and month 12
  M1/P1 et M1 / M2 angle measured just at the end of the intervention and at long time
12-month surgery rate | month 12
  use of surgery 12 months after randomization
Quality of life measured by the American Orthopedic Foot and Ankle Society score | day 0, day 75, month 6 and month 12
  American Orthopedic Foot and Ankle Society - hallux metatarsophalangeal interphalangeal scale (min = 0, max = 100, higher scores mean a better outcome).
Quality of life measured by the Foot Function Index score | day 0, day 75, month 6 and month 12
  Foot Fonction Index (min = 0, max = 100, higher scores mean a worse outcome).
Quality of life measured by the EuroQol Visual Analogue Scale | day 0, day 75, month 6 and month 12
  EuroQol Visual Analogue Scale (min = 0, max = 100, higher scores mean a better outcome.
Pain Visual Analogue Scale | day 0, day 75, month 6 and month 12
  Pain Visual Analogue Scale (min = 0, max = 10, higher scores mean a worse outcome).
Physician clinical qualitative assessement of skin condition | day 0 and day 75
  Presence or absence of irritation, blisters, redness, itching

CONTACTS AND LOCATIONS:
Overall Officials: Guy Allamel, PhD, Principal Investigator — CH Annecy Genevois
Locations (1):
- Centre Hospitalier Annecy Genevois, Metz-Tessy, France